CLINICAL TRIAL: NCT02231021
Title: Multicenter, Randomized, Double Blind, Three-arm Parallel Group Study to Evaluate Efficacy and Safety of Alogliptin and Pioglitazone Combination Therapy on Glucose Control in Type 2 Diabetes Subjects Who Have Inadequate Control With Metformin Monotherapy in Korea
Brief Title: The Practical Evidence of Antidiabetic Combination Therapy in Korea
Acronym: PEAK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kun-Ho Yoon (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor-Investigator, Kun-Ho Yoon, Professor, The Catholic University of Korea
Organization: The Catholic University of Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALO-IIT-012
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 2; alogliptin; pioglitazone; DPP4 inhibitor; thiazolidinedione
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — alogliptin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- alogliptin + pioglitazone (Experimental): alogliptin 25 mg 1 tablet daily for 24 weeks pioglitazone 30 mg 1 tablet daily for 24 weeks metformin for 24 weeks as the same dose and frequency as before enroll
  Interventions: Drug: alogliptin + pioglitazone
- alogliptin (Active Comparator): alogliptin 25 mg 1 tablet daily for 24 weeks pioglitazone matching placebo 1 tablet daily for 24 weeks metformin for 24 weeks as the same dose and frequency as before enroll
  Interventions: Drug: alogliptin
- Pioglitazone (Active Comparator): alogliptin matching placebo 1 tablet daily for 24 weeks pioglitazone 30 mg 1 tablet daily for 24 weeks metformin for 24 weeks as the same dose and frequency as before enroll
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: alogliptin — alogliptin 25 mg add-on background medication metformin
  Other Names: Nesina
  Arms: alogliptin
Drug: Pioglitazone — pioglitazone 30 mg add-on background medication metformin
  Other Names: actos
  Arms: Pioglitazone
Drug: alogliptin + pioglitazone — alogliptin 25 mg and pioglitazone 30 mg add-on background medication metformin
  Other Names: Nesina; Actos
  Arms: alogliptin + pioglitazone

SUMMARY:
This study evaluate the efficacy and safety of alogliptin and pioglitazone combination therapy in comparison with either alogliptin or pioglitazone on glucose control in the metformin-treated type 2 diabetic patients in Korea.

DETAILED DESCRIPTION:
Pathophysiology of type 2 diabetes is known as insulin resistance and progressive beta cell dysfunction.

Combination therapy with biguanides, glucagon-like peptide-1(GLP-1) agonists or dipeptidyl peptidase-4 inhibitor(DPP4I) and thiazolidinediones(TZD) seems reasonable theoretically, for their effects on different pathophysiologic defects.

Current treatment guidelines recommend a stepwise approach starting with lifestyle modification or lifestyle modification + metformin monotherapy, with recent focusing on patient individualization.

In Korea, Korean Diabetes Association also recommends stepwise approach and at the same time, emphasizes on the initial aggressive treatment including oral combination or insulin therapy according to HbA1c level to achieve target goal <6.5%.

Guide to the efficacy, timing, options of combination therapy is not clearly defined due to lack of sufficient evidences yet.

There is no clear report to demonstrate the clinical benefit of initial TZD and DPP4I combination therapy in the Korean.

Thus it is reasonable to study the effect of combination therapy in the patients with sub-optimal glucose control with metformin therapy only, comparing various combination options metformin with DPP4I only, TZD only, or both.

The hypothesis of this study is that combination therapy of alogliptin and pioglitazone added on the metformin has superior effect on HbA1c reduction than metformin and either alogliptin or pioglitazone in 6 month treatment.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the investigator, the subject is capable of understanding and complying with protocol requirements
* The subject or, when applicable, the subject's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures
* The subjects diagnosed type 2 diabetes mellitus at least 6 months
* Male and female and 19 to 75 years, inclusive
* 7.0% =<HbA1c =<10.0%
* 18.5 Kg/m2 =<Body Mass Index(BMI) =<45 kg/m2
* systolic/diastolic blood pressure =<160/100 at baseline
* hemoglobin of at least 12 g/dL for men and at least 10 g/dL for women
* A female subject of childbearing potential who is sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from singing of informed consent throughout the duration of the study
* Patient who receiving maximal tolerated dose of metformin at least 12 weeks without dose change (for metformin, >= 1,000 mg/day
* fasting c-peptide greater than 0.78 ng/mL(0.26 nmol/L) at baseline

Exclusion Criteria:

* The patient has received investigational compound(alogliptin or pioglitazone) within 180 days prior to baseline
* Patient who currently taking or need to take andy medicine which may exert a significant influence on blood glucose control except metformin.
* Severe renal disease : estimated glomerular filtration rate <50 mL/min
* Severe liver disease or AST, ALT >= 2.5 upper limit of normal
* Cardiac status : New York Heart Association III ~ IV
* Hypopituitarism or adrenal insufficiency
* Patient who has a history of major surgery, Severe infections, Severe traumas within 6 months
* Patients who has diagnosed malignancy within 5yrs ,
* Patients with active bladder cancer
* Patient with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
* Patient who has a history of hypersensitivity to Alogliptin, Pioglitazone or their ingredients
* Pregnant or lactating woman
* Patient who has history of excessive alcohol abuse
* Subject who is involved in other clinical trial within 90 days prior to initiation of this study.
* Subject who the investigator deems inappropriate to participate in this study

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Change in glycohemoglobin(HbA1c) from baseline | baseline, 24 weeks

SECONDARY OUTCOMES:
Proportion of subjects achieving HbA1c < 7.0% | 24 week
Proportion of subjects achieving HbA1c <6.5% | 24 week
Changes in glycated albumin(GA) from baseline | baseline, 24 weeks
Change in GA/HbA1c ratio from baseline | baseline, 24 weeks
Change in fasting blood sugar from baseline | baseline, 24 weeks
Incidence of hyperglycemic rescue | 12 week
  at Week 12, HbA1c >9.0%
Change in HbA1c from baseline | 12 week
Change in total cholesterol from baseline | baseline, 24 weeks
Change in triglycerides from baseline | baseline, 24 weeks
Change in LDL-cholesterol from baseline | baseline, 24 weeks
Change in HDL-cholesterol from baseline | baseline, 24 weeks
Changes in glycated albumin(GA) from baseline | baseline, 12 weeks
Change in GA/HbA1c ratio from baseline | baseline, 12 weeks
Change in fasting blood sugar from baseline | baseline, 12 weeks
Change in total cholesterol from baseline | baseline, 12 weeks
Change in triglycerides from baseline | baseline, 12 weeks
Change in LDL-cholesterol from baseline | baseline, 12 weeks
Change in HDL-cholesterol from baseline | baseline, 12 weeks
Change in Homeostasis Model Assessment-Insulin resistance(HOMA-IR) from baseline | baseline, 24 weeks
  a marker of insulin resistance
Change in Homeostasis Model Assessment - beta cell (HOMA-beta) from baseline | baseline, 24 weeks
  a marker of beta cell function
Change in highly sensitive C reactive protein(hs-CRP) from baseline | baseline, 24 weeks
  a marker of inflammation
Change in Plasmonogen activator inhibitor-1(PAI-1) from baseline | baseline, 24 weeks
Change in B-type natriuretic pepetide(BNP) from baseline | baseline, 24 weeks
event rate of hypoglycemia | upto 24 weeks
  A number of total event of hypoglycemia defined as blood glucose <70mg/dL or subjective symptom of typical hypoglycemia
No of subject with adverse event of special interest | upto 24 weeks
  The event of special interest include
  * heart failure
  * cardiovascular effect other than heart failure
  * edema
  * weight gain
  * urinary bladder tumor
  * macular edema
  * fracture of bone
  * pancreatitis
The number of serious adverse events | upto 24 weeks
The number of subject with hypersensitivity to study drugs | upto 24 weeks
The number of subject with any abnormality of laboratory evaluation | 12 week
  * Complete Blood count
  * BUN, Creatinine, AST, ALT, Calcium, Phosphorous, Sodium, Potassium, Total Protein, Albumin, Total Bilirubin, Gamma-glutamyl transferase, Alkaline phosphatase, Creatinine Kinase, amylase, lipase
  * Urine analysis including microscopic examination
The number of subject with any abnormality of laboratory evaluation | 24 week
  * Complete Blood count
  * Blood urea nigrogen, Creatinine, Aspartate aminotransferase, Alanine Aminotransferase, Calcium, Phosphorous, Sodium, Potassium, Total Protein, Albumin, Total Bilirubin, Gamma-glutamyl transferase, Alkaline phosphatase, Creatinine Kinase, amylase, lipase
  * Urine analysis including microscopic examination
The number of subject with any change of findings in Chest X-ray from baseline | 24 week
The number of subject with any change of findings in electrocardiogram from baseline | 24 week

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ho Yoon, MD, PhD, Principal Investigator — Seoul St Mary's Hospital, The Catholic Univerisity of Korea
Locations (1):
- Seoul St Mary's Hospital, The Catholic University of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No